CLINICAL TRIAL: NCT05662956
Title: Venetoclax/Azacitidine/Low-Dose Cytarabine/Aclarubicin/G-CSF (VA-CAG) in Newly-Diagnosed Acute Myeloid Leukemia: A Phase-2, Multi-center, Prospective Clinical Study
Brief Title: A Clinical Study of VA-CAG as Induction Therapy in Newly Diagnosed AML Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hematology department of the 920th hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMHD-01
Record Dates: First submitted 2022-12-10; First posted 2022-12-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Venetoclax; Azacitidine; Granulocyte colony-stimulating factor(G-CSF); Cytarabine; Aclarubicin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Induction: Subjects who meet the enrollment conditions will receive Venetoclax plus Azacitidine and CAG(VA-CAG) . Participants will receive this induction Therapy as azacitidine on days 1-7, venetoclax aily on days 1-28, cytarabine q12h on days 1-7, aclacinomycin on days 1,3,5,7, and granulocyte colony-stimulating factor on days 0-8. Participants will receive second induction if not reach complete remission.
  Consolidation: If patients are intermediate or poor risk and have plans for allogeneic hematopoietic stem-cell transplantation(allo-HSCT) , high dose cytarabine (3g/m2 q12h days 1-3) for 1-2 cycles and follow up with allo-HSCT. In other cases, high dose cytarabine for 4 cycles.
  Interventions: Drug: Venetoclax in combination with azacitidine and CAG

INTERVENTIONS:
Drug: Venetoclax in combination with azacitidine and CAG — Induction:
  VA regimen：
  Drug: Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-21);
  Drug: Azacitidine 75 mg/m2 subcutaneously once daily on days 1-7.
  CAG regimen：
  Drug: Cytarabine 10mg/m2 subcutaneously q12h on days 1-7;
  Drug: Aclacinomycin 12-14mg/m2 on days 1,3,5,7;
  Drug: Granulocyte colony-stimulating factor 5ug/kg on days 0-8, discontinue if WBC >20×10^9/L；
  Consolidation:
  Drug: Cytarabine 3g/m2 q12h on days 1-3.
  Other Names: VA-CAG regimen

SUMMARY:
This study aims to assess the therapeutic efficacy and safety of venetoclax in combination with azacitidine and CAG(VA-CAG) as induction regimen in newly diagnosed young patients with acute myeloid leukemia(AML).

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II clinical trial to assess the therapeutic efficacy and safety of venetoclax in combination with azacitidine (VA) and CAG (G-CSF priming, low dose cytarabine, and aclarubicin) as induction regimen in newly diagnosed patients with acute myeloid leukemia (AML).

The combination of venetoclax and azacitidine is the standard therapy for elderly (> 60 year old) patients with newly diagnosed AML who are not eligible for intensive chemotherapy. Previous studies have shown that venetoclax plus intense chemotherapy represent promising efficacy in de novo AML patients with high complete remission rates and good tolerance. The preliminary results suggest that venetoclax in combination with azacitidine and CAG are well tolerated and effective for newly diagnosed young patients with AML. Thus, this phase II clinical trial is going to further explore its efficacy and safety. It is expected that about 100 patients will take part in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old and ≤ 65 years old
2. Newly diagnosed as AML patients according to 2016 World Health Organization (WHO) classification;
3. Patients without receiving prior therapy for AML;
4. Eastern Cooperative Oncology Group (ECOG) Performance status score less than 3;
5. Liver function: Total bilirubin ≦2 upper limit of normal (ULN); aspartate aminotransferase (AST) ≦3 ULN; alanine aminotransferase (ALT)≦3 ULN
6. Renal function：Ccr（Creatinine Clearance Rate） ≧30 ml/min; Scr (serum creatinine) ≦2 ULN
7. Heart function: left ventricular ejection fraction ≧45%
8. Patients must participate in this clinical trial voluntarily and sign an informed consent form.

Exclusion Criteria:

1. Acute promyeloid leukemia；
2. AML with central nervous system (CNS) infiltration；
3. Patients have received prior hypomethylating agents (HMA) therapy for myelodysplastic syndrome (MDS) and progressed to AML；
4. Patients with a life expectancy <3 months
5. Patients with uncontrolled active infection;
6. HIV infection;
7. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to: a) Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment; b) An active second cancer that requires treatment within 6 months of study entry.
8. Female who are pregnant, breast feeding or childbearing potential.
9. Patients deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
CR rate | At the end of Cycle 1 of induction (each cycle is about 30 days)

SECONDARY OUTCOMES:
Adverse Events | From the first day of induction until the starting day of the next cycle of therapy (up to 60 days）
  Safety and tolerability analysis will be assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Duration of remission | From the date of the first remission until the date of relapse (assessed up to 30 months)
  DOR was defined as the period from the time to acquire CR until relapse
Minimal Residual Disease negative remission rate (MRD-negative rate) | After 1 cycle of induction (each cycle is about 30 days)
  Percentage of participants who converted to MRD < 10^-3 by flow cytometry before initiation of consolidation therapy.

OTHER OUTCOMES:
Overall survival | From the first day of induction until the date of death from any cause, assessed up to 30 months
  Overall Survival will be defined as the time from administration of the initial doses until death from any cause.
Relapse-free survival | From the first day of induction until the date of relapse or the date of death from any cause, assessed up to 30 months
  Relapse-free survival will be defined as the time since date of CR until either relapse or death in remission.

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China